CLINICAL TRIAL: NCT00342277
Title: Microarray Expression Profiling to Identify Stereotypic mRNA Profiles in Human Parturition
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999056; OH99-CH-N056
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Preterm Birth; Premature Rupture of Membranes
Keywords: Genetic Risk Factors; Tissue Specific Expression; Quantitative Real Time PCR; Preterm Birth; Expression Profiling; Natural History
MeSH Terms: conditions — Premature Birth; Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pregnant Women: Consecutive pregnant women admitted with either: Preterm labor/delivery/PROM. Termdelivery without labor/spontaneous labor /chorioamnionitis/failed labor leading to c-section

SUMMARY:
The understanding of the biological mechanisms underlying preterm birth is very limited, making prevention of preterm birth difficult. The incidence of preterm birth worldwide varies between 6%-11% in singleton pregnancies, and 64-93% of preterm deliveries occur after the spontaneous onset of labor (preterm labor). The risk factors associated with preterm birth include demographic variables such as ethnic group, past obstetric history, and complications of the current pregnancy such as infection and fetal congenital anomalies. The current study aims to investigate the basic mechanisms of preterm labor by systematically cataloging the changes in expression levels of all expressed genes whose sequences are available. The goals will be accomplished by using microarray technology followed by subsequent confirmative or complementary analyses.

DETAILED DESCRIPTION:
The understanding of the biological mechanisms underlying preterm birth is very limited, making prevention of preterm birth difficult. The incidence of preterm birth worldwide varies between 6%-11% in singleton pregnancies, and 64-93% of preterm deliveries occur after the spontaneous onset of labor (preterm labor). The risk factors associated with preterm birth include demographic variables such as ethnic group, past obstetric history, and complications of the current pregnancy such as infection and fetal congenital anomalies. The current study aims to investigate the basic mechanisms of preterm labor by systematically cataloging the changes in expression levels of all expressed genes whose sequences are available. The goals will be accomplished by using microarray technology followed by subsequent confirmative or complementary analyses.

ELIGIBILITY:
* INCLUSION CRITERIA:

Consecutive patients admitted with the following diagnoses from four different ethnic groups (Hispanic, African American, Asian, and Caucasian):

1. Preterm labor with intact membranes and with

   1. acute inflammation;
   2. chronic villitis;
   3. vascular pathology;
   4. no identifiable lesions.
2. Preterm delivery without labor because of the following reasons:

   1. pre-eclampsia;
   2. abruptio placentae;
   3. fetal anomalies;
   4. Other complications (e.g. automobile accidents) that necessitate immediate delivery.
3. PROM leading to preterm delivery and with

   1. acute inflammation;
   2. chronic villitis;
   3. vascular pathology;
   4. no identifiable lesions.
4. Term delivery without labor and no identifiable lesions.
5. Term delivery in spontaneous labor and no identifiable lesions.
6. Term delivery with chorioamnionitis.
7. Term delivery with failed labor leading to ceasarean section.

EXCLUSION CRITERIA:

1. Refusal of written informed consent
2. Fetal or maternal conditions mandating immediate delivery (i.e. fetal distress, significant hemorrhage, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women aged 15 years and older at 18 - 36 weeks of gestation admitted with the following diagnoses:@@@1) preterm labor with intact membranes@@@2) preterm delivery without labor@@@3) PROM leading to preterm delivery@@@4) Term deliveries without labor/spontaneous labor/with chorioamnionitis/with failed labor leading to cesarean section
Sampling Method: Probability Sample
Enrollment: 6838 (Actual)
Dates: Start 1999-12-21 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
To identify genes that are up- or down-regulated in preterm delivery and preterm PROM using microarray expression profiling. | After the study is closed to accrual
  Investigate the basic mechanisms of preterm labor by systematically cataloging the changes in expression levels of all expressed genes whose sequences are available.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (4):
- Wayne State University, Detroit, Michigan, United States
- Sotero del Rio Hospital, Puente Alto, Chile
- Padova Hospital, Padua, Italy
- Seoul National University, Seoul, South Korea